CLINICAL TRIAL: NCT06496633
Title: Efficacy and Safety of Echocardiography-guided Percutaneous Intraventricular Septal Radiofrequency Ablation for Obstructive Hypertrophic Cardiomyopathy After Alcohol Septal Ablation
Brief Title: Echocardiography-guided Percutaneous Septal Radiofrequency Ablation for Obstructive HCM After Alcohol Septal Ablation
Acronym: HCM
Status: Active, not recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Liu Liwen, Ph.D, Xijing Hospital
Other Study IDs: KY20242206-C-1
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-03

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Percutaneous Intramyocardial Septal Radiofrequency Ablation; Hypertrophic Cardiomyopathy; Alcohol Septal Ablation
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — We collected 10 ml of peripheral venous blood from the HCM patient and extracted the genome from the isolated white blood cells using The Relax Gene Blood DNA System (cat. no. DP319; Tiangen Biotech Co, Ltd., Beijing, China). After gene extraction, 96 cardio-disease-related genes were analyzed by an experienced genetic Counselor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort :Hypertrophic Cardiomyopathy patients with residual obstruction after Alcohol Septal Ablation: All patients performed procedure of Percutaneous Intramyocardial Septal Radiofrequency Ablation
  Interventions: Procedure: Percutaneous Intramyocardial Septal Radiofrequency Ablation

INTERVENTIONS:
Procedure: Percutaneous Intramyocardial Septal Radiofrequency Ablation — PIMSRA procedure represents a significant breakthrough in the treatment of HOCM patients, as it uses a unique transmyocardial approach to directly and precisely insert a radiofrequency electrode needle into the hypertrophied IVS for targeted ablation

SUMMARY:
After alcohol ablation, some HOCM patients have serious clinical symptoms and adverse complications, and need to undergo invasive surgery again when adequate drug therapy is not effective or cannot tolerate the side effects of drugs. Liwen surgery is a safe and effective new minimally invasive treatment for HOCM patients, so the purpose of this study was to evaluate the safety and efficacy of Liwen surgery in HOCM patients who failed alcohol ablation and provide new treatment methods for patients.

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is the most common inherited cardiovascular disease, mostly due to mutations in the gene encoding myocardial sarcomere contractile protein, with an incidence of about 1:500-1:200. HCM is the main cause of sudden cardiac death in young people and athletes. Its clinical manifestations are highly heterogeneous. Some patients have no obvious symptoms or mild symptoms, but some patients have obvious myocardial hypertrophy in the early stage, resulting in chest tightness, chest pain, breathing difficulties, syncope, heart failure, and even sudden cardiac death. The annual mortality rate of HCM patients is about 1.4% -2.2%. Alcohol septal ablation (ASA) is a kind of interventional therapy. Its principle is to inject anhydrous alcohol through a catheter, occlude the septal branch of the coronary artery, make the hypertrophic ventricular septal myocardium that dominates it ischemic, necrosis, thinning, and contractility decrease, so that the obstruction of the outflow tract disappears or alleviates, thereby improving the clinical symptoms of patients. However, HOCM patients often have serious clinical symptoms and adverse complications after alcohol ablation, and invasive surgical treatment is required when adequate drug therapy is not effective or cannot tolerate the side effects of drugs. Liwen surgery is a safe and effective new path to treat minimally invasive HOCM patients, so the purpose of this study was to evaluate the safety and efficacy of Liwen surgery after alcohol ablation in HOCM patients, and to verify its early postoperative efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is at least 18 years of age.
2. Hypertrophic cardiomyopathy with alcohol ablation, LVOT pressure difference at rest or after excitation ≥ 50mmHg;
3. The clinical symptoms are obvious, fatigue, shortness of breath, exhaustive angina pectoris, syncope, etc. seriously affect the quality of life, and the effect of adequate drug treatment is not good or the side effects of drugs cannot be tolerated;
4. After the informed consent of the patient and his family, he voluntarily underwent Liwen surgery.

Exclusion Criteria:

1. Non-obstructive hypertrophic cardiomyopathy;
2. Left ventricular hypertrophy due to secondary causes, such as increased preload, history of taking drugs suspected of causing left ventricular hypertrophy, etc.
3. Preoperative complications with other heart diseases require surgical treatment.
4. The disease will make it difficult to evaluate treatment (e.g. cancer, severe metabolic diseases, mental illness, etc.).
5. Patients who have participated in any clinical trial of drugs and/or medical devices within 1 month before surgery or during follow-up;
6. Pregnant and breastfeeding women;
7. Patients with poor adherence may not cooperate during treatment or follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with obstructive hypertrophic cardiomyopathy who underwent Liwen surgery at the Multidisciplinary Diagnosis and Treatment and Genetic Counseling Center for Hypertrophic Cardiomyopathy at Xijing Hospital of the Air Force Military Medical University from January 2017 to August 2023, all of whom had a history of alcohol ablation
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
treatment success rate | Six months after procedure.
  For survival, the left ventricular outflow tract pressure gradient (LVOT pressure gradient) decreased by ≥ 50% or the resting left ventricular outflow tract pressure gradient (LVOT pressure gradient) was < 30 mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Ultrasonic Diagnosis Department of Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Zhang J, Hsi DH, Ta S, Wang J, Wang B, Ma H, Shan B, Hu R, Li J, Liu L. Percutaneous Intramyocardial Septal Radiofrequency Ablation for Hypertrophic Cardiomyopathy With Residual Obstruction After Alcohol Septal Ablation. Can J Cardiol. 2025 Dec;41(12):2397-2406. doi: 10.1016/j.cjca.2025.08.355. Epub 2025 Sep 25. PMID 41015247